CLINICAL TRIAL: NCT03475810
Title: The Effect of Virtual Reality Glasses on Anxiety During Surgery Under Spinal Anesthesia: A Randomize Controlled Study
Brief Title: The Effect of Virtual Reality Glasses on Anxiety During Surgery Under Spinal Anesthesia
Acronym: VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ayse Zeynep Turan, Principle Investigator, Derince Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DerinceTRH-02
Record Dates: First submitted 2018-03-17; First posted 2018-03-23 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: VIRTUAL REALITY
Keywords: VIRTUAL REALITY; ANXIETY; SPINAL ANESTHESIA
MeSH Terms: conditions — Anxiety Disorders | interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR GROUP (Experimental): Patients watches 3D documentary videos on virtual reality glasses
  Interventions: Device: Virtual Reality; Drug: Midazolam
- midazolam (Active Comparator): Patients do not watch virtual reality videos but will be administered iv sedative drugs before spinal attempt.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Device: Virtual Reality — Patients will wear virtual reality glasses and start watching 3 D video after confirmation of adequate motor and sensorial block.
  Other Names: VR
  Arms: VR GROUP
Drug: Midazolam — 1-2 mg midazolam will be administered before spinal punction performed.
  Other Names: Demizolam

SUMMARY:
The aim of the study is to evaluate the efficacy of virtual reality glasses on anxiety of the patients who underwent operations under spinal anesthesia during peroperative period. Both control group and VR group will be carry out STAI- Traıt anxiety test before operation and trait test after operation. Patients will be perform spinal anesthesia after standard sedation administration. After block reach adequate level for operation patients in VR group will wear the glasses and started to watch a documentary about birds and a sedative music by the headset. Patients in Control group will take standard anesthesia care. Hemodynamic changes (systemic blood pressure, heart rate, respiration rate and pSPO2) will be record in both groups.

DETAILED DESCRIPTION:
The ASA score I-III Patients undergoing operation in OR under spinal anesthesia will be included in the study. Patients randomly assigned to VR group or Control Group. Patients will be carry out STAI-Trait Anxiety test preoperatively and second STAI test postoperatively. Spinal anesthesia will be performed after standard iv midazolam administration in both groups. After block reach adequate level for operation patient will wear the glasses and started to watch a documentary about birds and a sedative music by the headset in VR group and patient will take standard anesthesia care in Control group. The hemodynamic variables will be recorded during operation.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Patients who undergo surgery under spinal anesthesia
* American Society of Anesthesiologists (ASA) physical status classification I-III

Exclusion Criteria:

* patients undergo urgent operations
* patients have psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
State Anxiety Test | postoperative 20th min.
  State Anxiety test will be perform at postop care unit

SECONDARY OUTCOMES:
Total tolerance time of Virtual Reality glasses | intraoperative
  Total tolerance to VR glasses will be recorded
incidence of vomiting | intraoperative
  incidence of vomiting due to VR glasses
incidence of nausea | intraoperative
  incidence of nausea due to VR glasses
incidence of dizziness | intraoperative
  incidence of dizziness due to VR glasses
incidence of headache | intraoperative
  incidence of headache due to VR glasses
Postoperative Visual Analog Scale Score | postoperative 20 th min.
  Patient will be asked his anxiety level by Visual analog scale (VAS) from 0 to 10. 0(= no anxiety), 10(= highest level of anxiety)
change in mean arterial pressure | 5th min. intraoperative
  blood pressure of the patient will be measured noninvasively from proper extremity in the operating room
change in mean arterial pressure | 10th min. intraoperative
  blood pressure of the patient will be measured noninvasively from proper extremity in the operating room
change in mean arterial pressure | 15th min. intraoperative
  blood pressure of the patient will be measured noninvasively from proper extremity in the operating room
change in mean arterial pressure | 20th min. intraoperative
  blood pressure of the patient will be measured noninvasively from proper extremity in the operating room
change in heart rate | 5th min. intraoperative
  heart rate of the patient will be monitored and recorded
change in heart rate | 10th min. intraoperative
  heart rate of the patient will be monitored and recorded
change in heart rate | 15th min. intraoperative
  heart rate of the patient will be monitored and recorded
change in heart rate | 20th min. intraoperative
  heart rate of the patient will be monitored and recorded
change in respiratory rate | 5th min. intraoperative
  respiratory rate of the patient will be monitored and recorded
change in respiratory rate | 10th min. intraoperative
  respiratory rate of the patient will be monitored and recorded
change in respiratory rate | 15th min. intraoperative
  respiratory rate of the patient will be monitored and recorded
change in respiratory rate | 20th min. intraoperative
  respiratory rate of the patient will be monitored and recorded

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Zeynep Turan, MD, Principal Investigator — Derince Research and Training Hospital
Locations (1):
- Derince Research and Training Hospital, Kocaeli, Turkey (Türkiye)